CLINICAL TRIAL: NCT02850471
Title: Pulmonary Protection of Transcutaneous Electrical Acupoint Stimulation in Gynecologic Laparoscopic Surgery
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: we need more participants to complete the research
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Yanchao Yang, resident doctor, Shengjing Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: pulmonary protection
Record Dates: First submitted 2016-07-21; First posted 2016-08-01 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-07

CONDITIONS: Reperfusion Injury
Keywords: Postoperative pulmonary complications; Transcutaneous electric acupoint stimulation; pulmonary protection
MeSH Terms: conditions — Reperfusion Injury | interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TEAS group (Experimental): Before anesthesia, patients in this group treated with Transcutaneous Electric Acupoint Stimulation (TEAS) which is an electroacupuncture on Feishu, Hegu, Chize half an hour before the surgery, using the device Hua Tuo SDZ-II Acupoint Stimulator. The stimulus parameters set as 2/100Hz, 2V, 30min.
  Interventions: Device: electroacupuncture
- controlled group (No Intervention): Patients in controlled group treated without TEAS or other placebo.

INTERVENTIONS:
Device: electroacupuncture — Transcutaneous Electric Acupoint Stimulation which is a device of electroacupuncture was used on patients in TEAS group with the stimulator parameters set as 2/100Hz, 2V, 30min.
  Arms: TEAS group

SUMMARY:
TEAS might protect against postoperative pulmonary such as ischemia-reperfusion injury (IRI) and atelectasis. We tested the hypothesis that transcutaneous electrical acupoint stimulation protects against postoperative pulmonary complications in patients who are receiving mechanical ventilation during general anesthesia for gynecologic laparoscopic surgery.

DETAILED DESCRIPTION:
Participants: 100 patients who underwent elective gynecologic laparoscopic surgery Methods: We recruited 100 patients who are planned for gynecologic laparoscopic surgery. Patients were enrolled from March 1, 2015. We randomly allocated patients into two groups: controlled group ( patients treated without transcutaneous electrical acupoint stimulation) and TEAS group (patients treated with TEAS on Feishu, Hegu, Chize half an hour before the surgery). Blood pH, Pco2, Po2 and oxygen saturation were measured by an automatic blood gas analyzer immediately after obtaining the samples from the aorta. Sample all the patients blood before and after the surgery. And then measure the level of TNF-α, IL-1β, and IL-6.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 65 to 75
* The American Society of anesthesiologists (American Society of Anesthesiology, ASA) class Ⅱ ~ III
* scheduled for gynecologic laparoscopic surgery under general anesthesia

Exclusion Criteria:

* pre-existing lung or caridac disease
* impaired kidney or liver function
* history of bronchial asthma or chronic obstructive pulmonary disease
* history of smoking
* respiratory infection in the previous 2 weeks
* preoperative use of bronchodilator, or a steroid

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-03; Primary Completion 2015-12 (Actual); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
the change of hemodynamic parameter MAP in mmHg | intraoperative
the change of hemodynamic parameters HR in beat per minutes | intraoperative
the change of blood SPO2 in percentage | intraoperative
the change of blood pH | intraoperative
the change of blood PCO2 in mmHg | intraoperative
the change of blood PO2 in mmHg | intraoperative

SECONDARY OUTCOMES:
the change of Plasma concentration of TNF-α in pg/mL | intraoperative
post-operative pulmonary complications | in the first 5 days after surgery
the change of plasma concentration of IL-1β | intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: Junchao Zhu, doctor, Study Director — professor
Locations (1):
- Shengjing hospital of China medical university, Shenyang, Liaoning, China

REFERENCES:
- [Derived] Wei W, Bai W, Yang Y, Li Y, Teng X, Wan Y, Zhu J. Pulmonary protection of transcutaneous electrical acupoint stimulation in gynecological laparoscopic surgery: A randomized controlled trial. Exp Ther Med. 2020 Jan;19(1):511-518. doi: 10.3892/etm.2019.8245. Epub 2019 Nov 26. PMID 31885697